CLINICAL TRIAL: NCT06385548
Title: Phase I-II Study to Evaluate the Safety, Tolerability, and Efficacy of Lurbinectedin and Dostarlimab in Patients with Advanced/Recurrent Endometrial Cancer with Disease Progression Following Previous Platinum Chemotherapy Therapy
Brief Title: Efficacy and Safety Study of Lurbinectedin and Dostarlimab in Cancer Patients: Protocol VHIO21001 - LiDer
Acronym: LiDer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IMP owner decision
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHIO21001
Record Dates: First submitted 2024-04-11; First posted 2024-04-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; lurbinectedin; dostarlimab
MeSH Terms: conditions — Endometrial Neoplasms | interventions — PM 01183; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lurbinectedin and Dostarlimab Combination Therapy (Experimental)
  Interventions: Drug: Lurbinectedin; Drug: Dostarlimab

INTERVENTIONS:
Drug: Lurbinectedin — participants will receive intravenous infusions of lurbinectedin at a dose of 2.6 mg/m², diluted in a minimum of 100 mL of either 5% glucose solution or 0.9% sodium chloride solution. The infusion will last for one hour and will be administered every three weeks.
Drug: Dostarlimab — participants will receive intravenous infusions of dostarlimab at a fixed dose of 500 mg, administered over 30 minutes on Day 1 of each three-week cycle.

SUMMARY:
Background:

Endometrial cancer is a prevalent gynecological malignancy, with a significant number of cases diagnosed at an advanced stage or recurring following initial treatment. Platinum-based chemotherapy represents a standard treatment option for these patients; however, disease progression often occurs, highlighting the need for novel therapeutic approaches. Lurbinectedin, a synthetic analog of marine alkaloid-derived compounds, and dostarlimab, a monoclonal antibody targeting PD-1, have demonstrated promising antitumor activity in various malignancies. This phase I-II clinical trial seeks to evaluate the safety, tolerability, and efficacy of combining lurbinectedin and dostarlimab in patients with advanced or recurrent endometrial cancer who have experienced disease progression following platinum-based chemotherapy.

Primary Objectives:

To determine the maximum tolerated dose (MTD) and recommended dose for further investigation of lurbinectedin and dostarlimab in combination therapy for advanced or recurrent endometrial cancer.

To assess the antitumor activity of lurbinectedin and dostarlimab combination therapy, measured by objective response rate (ORR), in patients with advanced or recurrent endometrial cancer.

Secondary Objectives:

To evaluate the safety and tolerability of lurbinectedin and dostarlimab combination therapy in patients with advanced or recurrent endometrial cancer.

To characterize the pharmacokinetic profile of lurbinectedin and dostarlimab when administered in combination therapy.

To explore pharmacogenomic biomarkers predictive of response and/or resistance to lurbinectedin and dostarlimab combination therapy in patients with advanced or recurrent endometrial cancer.

To assess progression-free survival (PFS), duration of response (DOR), clinical benefit rate (CBR), and overall survival (OS) in patients receiving lurbinectedin and dostarlimab combination therapy for advanced or recurrent endometrial cancer.

To investigate the impact of lurbinectedin and dostarlimab combination therapy on quality of life and symptom control in patients with advanced or recurrent endometrial cancer.

DETAILED DESCRIPTION:
This study is a phase I-II clinical trial conducted to evaluate the safety, tolerability, and efficacy of lurbinectedin and dostarlimab combination therapy in patients with advanced or recurrent endometrial cancer. The trial follows a multicenter, open-label design and comprises two phases: a dose escalation phase (Phase I) and an expansion phase (Phase II). The primary endpoints include determining the maximum tolerated dose (MTD), recommended dose for further investigation, and objective response rate (ORR). Secondary endpoints encompass safety, pharmacokinetics, pharmacogenomics, progression-free survival (PFS), duration of response (DOR), clinical benefit rate (CBR), overall survival (OS), and quality of life assessments.

Study Treatments:

Lurbinectedin: Lurbinectedin is administered as a lyophilized powder for concentrate for infusion, reconstituted with sterile water for injection to achieve a concentration of 0.5 mg/mL. The initial dose for infusion is 2.6 mg/m^2, diluted in either 5% glucose solution or 0.9% sodium chloride solution. During Phase I, dose adjustments are based on body surface area calculated using the DuBois formula.

Dostarlimab: Dostarlimab is supplied in vials containing 500 mg at a concentration of 50 mg/mL. The recommended dose is a fixed dose of 500 mg administered intravenously over 30 minutes. Treatment cycles consist of administration on Day 1 of a 21-day cycle, with dostarlimab followed by lurbinectedin in combination therapy.

During the dose escalation phase (Phase I), a predefined dose escalation scheme is employed, starting with dose level (DL) -1 and progressing to DL1, DL2, and subsequent levels as per the protocol. Dose escalation is guided by the occurrence of dose-limiting toxicities (DLTs) and the determination of the MTD. Once the MTD is established, the expansion phase (Phase II) begins, wherein additional patients receive treatment at the recommended dose to further evaluate safety and efficacy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Histologically confirmed advanced or recurrent endometrial cancer.
* Disease progression following prior platinum-based chemotherapy.
* Adequate organ function, including bone marrow, renal, and hepatic function.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Measurable disease per RECIST v.1.1 criteria.
* Availability of archival tumor tissue sample or willingness to undergo a tumor biopsy.
* Signed informed consent form.
* Life expectancy of at least 3 months.
* Willingness and ability to comply with study procedures and follow-up visits.
* Agreement to use effective contraception during the study period and for a specified duration thereafter if applicable.

Exclusion Criteria:

* Prior treatment with lurbinectedin or dostarlimab.
* Active autoimmune disease requiring systemic treatment.
* Symptomatic or untreated central nervous system metastases.
* History of interstitial lung disease or pneumonitis requiring steroids.
* Uncontrolled concurrent illness or medical condition.
* History of Grade ≥3 immune-related adverse events with prior immunotherapy.
* Pregnancy or breastfeeding.
* Concurrent treatment with other anticancer therapy.
* Prior treatment with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Concurrent treatment with corticosteroids exceeding a specified dose or duration.
* Participation in another clinical trial involving investigational therapy within a specified timeframe.
* Any other condition that, in the investigator's opinion, would compromise the patient's safety or interfere with the study conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-05-01 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Dose (RD) Determination | MTD and RD will be assessed during the Phase I portion of the study, the time frame will be arround 6 months.
  This measure involves identifying the highest dose of lurbinectedin in combination with dostarlimab that can be administered without causing unacceptable toxicity. The recommended dose for further evaluation in Phase II will also be determined.
Evaluation of Lurbinectedin and Dostarlimab Combination Therapy in Advanced/Recurrent Cervical Cancer Patients | This objective will be assessed during the Phase II portion of the study, the time frame will be arround 6 months.
  This objective aims to assess the efficacy of lurbinectedin in combination with dostarlimab in advanced or recurrent cervical cancer patients who have experienced disease progression after platinum-based chemotherapy. The primary objective is to evaluate the confirmed tumor response rate, as defined by RECIST v1.1 criteria, in patients without alterations in the MMR system.

SECONDARY OUTCOMES:
Safety Evaluation of Lurbinectedin in combination with Dostarlimab | Safety evaluations will occur throughout the study, starting from the first dose administration and continuing until the end of the study, an average of 1 year
  Safety will be assessed by monitoring adverse events (AEs) using the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
Evaluate the progression-free survival (PFS) | These efficacy endpoints will be evaluated throughout the study, with regular assessments during follow-up visits, up to 1 year
  Evaluate the time from study entry until disease progression or death from any cause.
Pharmacokinetic (PK) and Pharmacogenomic Evaluation | PK and pharmacogenomic evaluations will occur at specified time points during the study (12 months).
  PK parameters will be assessed to determine the drug's concentration in plasma over time.
Overall Response Rate (ORR) | ORR will be assessed after completion of treatment cycles and response evaluations according to RECIST v.1.1 criteria(1 year).
  The proportion of patients with a complete or partial response to treatment, assessed by RECIST v.1.1 criteria, specifically in the Phase II portion of the study.
Evaluate the Duration of Response (DOR) | Safety evaluations will occur throughout the study, starting from the first dose administration and continuing until the end of the study, an average of 1 year
  The objective is to analyse the time from the first documented response until disease progression or death.
Evaluate the Clinical Benefit Rate (CBR) | Safety evaluations will occur throughout the study, starting from the first dose administration and continuing until the end of the study, an average of 24 months
  The objective is to examinate the time from study entry until death from any cause. Survival Rates: The percentage of patients who survive at specified time points (6, 12, 18, and 24 months)

IPD SHARING:
Plan to Share IPD: No